CLINICAL TRIAL: NCT02001233
Title: An Open-labelled, Multicentered, Follow-up Study for a Phase III, Efficacy Trial to Evaluate the Two-year Efficacy, Safety, and Immune Persisitence of Inactivated Enterovirus Type 71 (EV71) Vaccine
Brief Title: A Follow-up Study for a Phase III, Efficacy Trial in Inactivated Enterovirus Type 71 (EV71) Vaccine
Status: Completed | Type: Observational
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-EV71-3003-0
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2022-05-26 (Actual); Status verified 2015-05

CONDITIONS: Hand, Foot and Mouth Disease
Keywords: EV71 vaccine; EV71-associated HFMD; efficacy; safety; immune persistence
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples will be taken from 1200 subjects in the immunogenicity subgroup 26 months after the first vaccination.
  Throat and anal swab samples will be taken from the cases with Hand, Foot and mouth disease for the detection of PCR assays and the isolation of EV71.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- EV71 Vaccine: Inactivated vaccine (vero cell) against EV71 of 400U /0.5ml in 5000 infants aged 6-35 months old on day0,28
  Interventions: Biological: EV71 vaccine
- Placebo: placebo in 5000 infants aged 6-35 months old on day0,28

INTERVENTIONS:
Biological: EV71 vaccine — inactivated vaccine (vero cell) against EV71 of 400U /0.5ml, two doses, 28 days interval
  Groups: EV71 Vaccine

SUMMARY:
The purpose of this follow-up study is to evaluate the two-year efficacy, immunogenicity and safety of EV71 Vaccines in preventing Hand, Foot and Mouth disease caused by EV71 in a total 10,000 healthy infants volunteers aged from 6 to 35months old.

DETAILED DESCRIPTION:
The phase III, efficacy trial of inactivated vaccine (vero cell) against EV71 has completed on March 2013 in China. The data from the phase III study suggested that the inactivated EV71 vaccine had protection effects on healthy Chinese infants against Hand, Foot and Mouth disease caused by EV71 within one-year surveillance period, and had clinically acceptable safety and good one-year immune persistence.

This study is the phase III, open-labelled, follow-up research, in order to evaluate the two-year efficacy, safety and immune persistence.

ELIGIBILITY:
Inclusion Criteria:

* All subjects vaccinated at least one injection of EV71 vaccine or the placebo in the phase III efficacy trial.

Exclusion Criteria:

* subjects who refuse to continue in the study.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy Chinese infants aged 6 to 35 months old
Sampling Method: Probability Sample
Enrollment: 10077 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The incidence rate of Hand, Foot and Mouth disease caused by EV71 within the second year observation period after the second vaccination | Within the second year after the second vaccination
  to evaluate the efficacy of EV71 vacccine against HFMD caused by EV71

SECONDARY OUTCOMES:
The GMT of anti-EV71 antibodies in serum two years after second vaccination | 26 months after second vaccination
  to evaluate the immune persistence of anti-EV71 antibodies in serum
Frequency of serious adverse events (SAEs) with the second year after the second vaccination | within the second year after the second vaccination
  Frequency of serious adverse events in healthy infants during the oney-year follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Cai Zhu, BS, Principal Investigator — Jiangsu Center for Diseases Control and Prevention
Locations (3):
- China (3):
  - Ganyu, Lianyungang, Jiangsu
  - Taixing, Taizhou, Jiangsu
  - Sheyang, Yancheng, Jiangsu